CLINICAL TRIAL: NCT06881160
Title: Circulating Mi-RNA Associated With Disease Severity and Outcome in COVID-19 Patients
Brief Title: Mi-RNA and COVID-19
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, TINELLI GIOVANNI, Associate Professor of Vascular Surgery, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 3155
Record Dates: First submitted 2023-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood Plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mild Respiratory Failure Covid-19: Patients with Covid-19 and mild respiratory failure defined as PaO2/FiO2 201-300 mm Hg
  Interventions: Diagnostic Test: mi-RNA analysis
- Severe Respiratory Failure Covid-19: Patients with Covid-19 and severe respiratory failure defined as PaO2/FiO2 ≤100 mm Hg.
  Interventions: Diagnostic Test: mi-RNA analysis

INTERVENTIONS:
Diagnostic Test: mi-RNA analysis — To identify biomarkers that could predict the risk of a worsened COVID-19 disease progression.

SUMMARY:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), the cause of coronavirus disease 2019 (COVID-19), induces a spectrum of clinical conditions ranging from asymptomatic infection to life threatening severe disease, characterized by respiratory failure, shock and multi-organ dysfunction requiring admission in the intensive care unit (ICU).

The aim of the present study is to analyze miRNAs associated with SARS-CoV-2 infection, disease severity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* 18 years
* diagnosis of SARS-CoV-2 infection confirmed by molecular testing on nasopharyngeal swabs

Exclusion Criteria:

* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted at the Fondazione Policlinico Gemelli IRCCS hospital with Covid-19 were enrolled. Peripheral blood samples were collected at the time of hospital admission. Plasma were separated from whole blood by centrifugation for 15 min at 3.000 rpm at 4°C and stored at -80°C until processing
Sampling Method: Non-Probability Sample
Enrollment: 49 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Severity of Covid-19 | Through study completion, an average of 1 year
  Severity of the disease

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No